CLINICAL TRIAL: NCT06505473
Title: Effects of Music Combined With Cognitive Behavioral Therapy on Chronic Subjective Tinnitus and a Multi-Factor Analysis
Brief Title: Effects of Music Combined With CBT on Chronic Subjective Tinnitus
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-453-01
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Subjective Tinnitus; Sleep Disorder
Keywords: chronic subjective tinnitus; music therapy; cognitive behavioral therapy; neural mechanism
MeSH Terms: conditions — Tinnitus; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pre-operative results: pre-operative period test results, baseline data.
  Interventions: Behavioral: music-CBT
- post-operative results: post-operative period test results, review data.
- healthy control: Subjects with no tinnitus and matched baseline information

INTERVENTIONS:
Behavioral: music-CBT — notched relaxation music combined with personalized CBT
  Groups: pre-operative results

SUMMARY:
This study retrospectively analyzed the first and second visit data of chronic subjective tinnitus patients who received music combined with cognitive behavioral therapy in our hospital in recent years. Behavioral tests and tinnitus questionnaires, as well as sleep and depression scores, were used to analyze the therapeutic effects of this approach. EEG results were analyzed as a potential neurobiological marker to explore the neural mechanism of tinnitus symptom improvement.

DETAILED DESCRIPTION:
The subjects of this study were chronic subjective tinnitus patients and normal controls who were treated with music therapy combined with cognitive behavioral therapy (music-CBT) in the Department of Otolaryngology of Sun Yat-sen Memorial Hospital from December 2016 to March 2024 and who had completed re-examination. The pre- and post-music-CBT data of past patients who met our study conditions were collected for retrospective statistics. The complete sample data included medical history, pure tone audiometry, tinnitus matching, tinnitus questionnaires (Tinnitus Handicap Inventory, Visual Analog Scales, tinnitus Functional Index), sleep quality questionnaire (Pittsburgh Sleep Quality Index), and depression questionnaire (Hamilton Depression Scale -24 items). The resting state electroencephalogram (rs-EEG). Retrospective statistical analysis was conducted to determine the clinical efficacy and influencing factors of music-CBT for chronic subjective tinnitus at 3 months and long term. Finally, the neural mechanism of music-CBT for tinnitus treatment was analyzed based on rs-EEG results.

ELIGIBILITY:
Inclusion Criteria:

* adults aged between 18 and 60
* a total score of 18 or higher on THI
* a constant tinnitus that can be matched
* right-handed
* no significant medical or psychiatric conditions

Exclusion Criteria:

* intermittent, pulsating or objective tinnitus
* central nervous system disease
* cognitive impairment
* other contraindications for EEG testing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants involved in this study were patients admitted to Sun Yat-sen Memorial Hospital with chronic subjective tinnitus that had lasted for more than six months. They were all treated with Music-CBT for 3 months.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
pure tone audiometry | the exact 1 day of the first visit
  The air conductivity threshold of pure tone audiometry across the frequency range of 500-4000Hz is referred to as the pure tone average (PTA) for the tested ear
tinnitus loudness | the exact 1 day of the first visit and review visit, within 3 - 4.5 months
  Tinnitus loudness was calculated by the matched intensity subtracting the pure tone threshold at that frequency.
tinnitus handicap inventory (THI) | the exact 1 day of the first visit and review visit, within 3 - 4.5 months
  There were 25 items in the THI scale, divided into three subscales (functional, emotional, and catastrophic), and response choices consisted of "no" (0 points), "sometimes" (2 points), and "yes" (4 points). A higher score of THI indicateed more severe tinnitus.
tinnitus functional index (TFI) | the exact day of the first visit and review visit, within 3 - 4.5 months
  The TFI scale assessed tinnitus-related distress and severity. It contained 8 subscales. They were denoted as TFI-I (Intrusiveness) and TFI-SC (Sense of) control), TFI-C (Cognition), TFI-S (Sleep), TFI-A (Auditory), TFI-R (Relaxation), TFI-Q (Quality of life), TFI-E (Emotional) distress); A total of 25 items are included. Each item worthes 100 points. The average score of all items was recorded as the total TFI score (0-100). A higher score of TFI indicateed more severe tinnitus.
EEG functional connectivity and brain network characteristics | the exact 1 day of the first visit and review visit, within 3 - 4.5 months
  EEG signals were used to explore the activation of brain regions and remodeling of poor connections in the postoperative outcomes of conductive hearing loss patients accompanied by with tinnitus. Power spectral density calculation, traceability analysis, functional connection, microstate, clustering coefficient, feature path length, feature path intermediation, and isocompatibility coefficient were collected and then analyzed.

SECONDARY OUTCOMES:
visual analogue scale (VAS) | the exact 1 day of the first visit and review visit, within 3 - 4.5 months
  VAS scaled from 0 to 10. A score of 0 means that tinnitus has no impact on daily life, and a score of 10 means that tinnitus has an intolerable, fatal level of impact on daily life.
Pittsburgh sleep quality index (PSQI) | the exact 1 day of the first visit and review visit, within 3 - 4.5 months
  PSQI scale was compiled by Buysse et al in 1989 to assess the sleep quality of individuals in the last 1 month. The total score ranges from 0 to 21. A higher score indicates worse sleep quality in the past month.
Hamilton Depression Scale -24 items (HAMD-24) | the exact 1 day of the first visit and review visit, within 3 - 4.5 months
  The HAMD-24 was used to assess the degree of depression and emotional state in patients with chronic subjective tinnitus. The assessment included the emotional state and symptoms of autonomic nervous system disorders in the past week, and each question was scored according to the presence and severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Haidi Yang, master, Study Director — SunYatSunU2H

IPD SHARING:
Plan to Share IPD: No